CLINICAL TRIAL: NCT06906042
Title: Multimodal Cardiovascular and Hepatic Population Imaging
Acronym: ICONIC
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C24-17; 2024-A02188-39 (Other: ANSM ID-RCB)
Record Dates: First submitted 2024-12-10; First posted 2025-04-02 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers; Imaging Evaluation
Keywords: multimodal imaging; heart; liver; Constances cohort; population; Cardiac imaging; MRI; Aging; reference values
MeSH Terms: interventions — Independent Medical Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Biobank blood samples (16 ml) will be collected and stored as follows:.
  * Dry blood tubes (8ml) for the constitution of a serum collection, stored in aliquots.
  * EDTA blood tubes (8 ml) for the constitution of a plasma collection, stored in aliquots.
  * For subjects who consent to genetic analysis (no additional intake) and according to the informed consent, the EDTA tube will be kepted at the CRB ICAN for future DNA extraction for ICONIC or further research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Constances volunteers: The 2400 volunteers will be stratifed according to age in decades from 20 to 80 years of age and matched 1:1 male:female.
  Interventions: Radiation: Imaging examinations; Other: Paramedical examinations; Other: Medical examination; Other: Echocardiography

INTERVENTIONS:
Radiation: Imaging examinations — * Cardiovascular MRI
  * Hepatic MRI
  * Hepatic ultrasound
Other: Paramedical examinations — * Urinary pregnancy test for women of childbearing age.
  * Blood sample for cardiometabolism profiling
  * Blood samples for biobanking (according to the information and consent form)
  * Impedancemetry
  * AGE reader: combined non-invasive measurement of aging and accumulation of glycated proteins in the subcutaneous tissue will be performed with a CE-marked device.
Other: Medical examination — * Review of risk factors
  * Review of previous history
  * Recording of current medication (dci, dose, start date)
  * Recording of medication in the last 6 months and discontinued since (dci, dose, start date)
Other: Echocardiography — Echocardiography including: 12-lead digital ECG

SUMMARY:
Medical imaging is increasingly important for understanding diseases, detecting them early, and personalizing treatments. New imaging techniques, which can measure processes in the body without surgery, are opening the door to a more precise approach to medicine. Instead of relying on general probabilities, this technology allows us to analyze specific factors in a person's health, leading to better predictions and targeted treatments. One key challenge in medicine today is reducing "residual individual risk"-the remaining health risks that current treatments don't fully address. This involves understanding how factors like age, sex, genetics, and environment affect our health, particularly when it comes to conditions like heart and liver disease. By using imaging to distinguish between normal aging and disease, we can better assess individual health risks.

The current project will create a large collection of medical images linked with health data from a broad population across France. Using advanced, non-invasive techniques such as MRI and ultrasound, researchers will analyze the heart, blood vessels, and liver in detail, considering factors like gender and health risk profiles. This will help improve our understanding of these diseases, which are often silent and not well understood, providing direct benefits to the participants. Ultimately, the goal is to optimize imaging technologies for large-scale studies, which will help enhance early detection and prevention for everyone.

ELIGIBILITY:
Inclusion Criteria:

* Participation to the Constances cohort
* Age ≥ 20 years
* No overt cardiovascular or hepatic disease or related symptoms
* No known family or personal genetic disease
* Affiliation with a social security scheme or beneficiary of such a scheme.
* Agreement to sign the consent

Exclusion Criteria:

* Renal function impairment with GFR < 60 mL/min/1.73m2
* Deprived of liberty or persons subject to a legal protection measure (under guardianship or trusteeship)
* People with contraindications to MRI (claustrophobia, presence of metallic elements…)
* Pregnant or breastfeeding woman (pregnancy urinary test before inclusion for women of childbearing age).

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants are asymptomatic volunteers from the Constances cohort, whose risk factor profiles are representative of the population in the Île-de-France region (Paris area). Participants are divided into 6 decades from 20 to 80 years with equal distribution of men/women (200 men and 200 women per decade)
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2030-03-14 (Estimated); Study Completion 2033-03-14 (Estimated)

PRIMARY OUTCOMES:
Establishement of reference nomograms accounting for age in heart | During 36 months of analysis (after 60 months of inclusion)
  Ultrasound and MRI images analysis of qualitative and quantitative morphology, function, quantitative tissue characterization of the heart
Establishement of reference nomograms accounting for sex in heart | During 36 months of analysis (after 60 months of inclusion)
  Ultrasound and MRI images analysis of qualitative and quantitative morphology, function, quantitative tissue characterization of the heart
Establishement of reference nomograms accounting for age in liver | During 36 months of analysis (after 60 months of inclusion)
  Ultrasound and MRI images analysis of quantitative steatosis, fibrosis
Establishement of reference nomograms accounting for sex in liver | During 36 months of analysis (after 60 months of inclusion)
  Ultrasound and MRI images analysis of quantitative steatosis, fibrosis
Establishement of reference nomograms accounting for age in adipose tissue | During 36 months of analysis (after 60 months of inclusion)
  Ultrasound and MRI images analysis of volumes of subcutaneous, visceral and epicardial adipose tissues
Establishement of reference nomograms accounting for sex in adipose tissue | During 36 months of analysis (after 60 months of inclusion)
  Ultrasound and MRI images analysis of volumes of subcutaneous, visceral and epicardial adipose tissues

SECONDARY OUTCOMES:
Advanced Imaging profiling of Heart | During 36 months of analysis (after 60 months of inclusion)
  Analysis of the cardiac cavities in 2D, 3D and in deformation by echocardiography analysis
Advanced imaging profiling in Liver | During 36 months of analysis (after 60 months of inclusion)
  Qualitative analysis of liver morphology and the nodularity of its boundaries, presence of ascites and portal derivation. Also presence of incidentaloma.
Advanced biological phenotyping | During 36 months of analysis (after 60 months of inclusion)
  Study of metabolic pathways and candidate biomarker suspected to be involved in aging
identification of genetic risk markers for cardio-metabolic diseases | During 36 months of analysis (after 60 months of inclusion)
  Defining the minimum set of markers useful for creating a risk score

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mauger CA, Gilbert K, Suinesiaputra A, Bluemke DA, Wu CO, Lima JAC, Young AA, Ambale-Venkatesh B. Multi-Ethnic Study of Atherosclerosis: Relationship between Left Ventricular Shape at Cardiac MRI and 10-year Outcomes. Radiology. 2023 Feb;306(2):e220122. doi: 10.1148/radiol.220122. Epub 2022 Sep 20. PMID 36125376
- [Result] Bohnen S, Avanesov M, Jagodzinski A, Schnabel RB, Zeller T, Karakas M, Schneider J, Tahir E, Cavus E, Spink C, Radunski UK, Ojeda F, Adam G, Blankenberg S, Lund GK, Muellerleile K. Cardiovascular magnetic resonance imaging in the prospective, population-based, Hamburg City Health cohort study: objectives and design. J Cardiovasc Magn Reson. 2018 Sep 24;20(1):68. doi: 10.1186/s12968-018-0490-7. PMID 30244673
- [Result] Nie C, Li Y, Li R, Yan Y, Zhang D, Li T, Li Z, Sun Y, Zhen H, Ding J, Wan Z, Gong J, Shi Y, Huang Z, Wu Y, Cai K, Zong Y, Wang Z, Wang R, Jian M, Jin X, Wang J, Yang H, Han JJ, Zhang X, Franceschi C, Kennedy BK, Xu X. Distinct biological ages of organs and systems identified from a multi-omics study. Cell Rep. 2022 Mar 8;38(10):110459. doi: 10.1016/j.celrep.2022.110459. PMID 35263580
- [Result] Laurent S, Boutouyrie P, Cunha PG, Lacolley P, Nilsson PM. Concept of Extremes in Vascular Aging. Hypertension. 2019 Aug;74(2):218-228. doi: 10.1161/HYPERTENSIONAHA.119.12655. Epub 2019 Jun 17. No abstract available. PMID 31203728